CLINICAL TRIAL: NCT01857752
Title: Phase II Study Temozolomide for Retinoblastoma Metastatic to the Central Nervous System for Patients From Guatemala
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: accrual
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEDSEYE0003; 22753 (Other: Stanford IRB)
Record Dates: First submitted 2013-03-25; First posted 2013-05-20 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Temozolomide

ARMS (1):
- temozolomide (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide

SUMMARY:
Primary Objectives:

1. To investigate the response rate (complete response plus partial response) of temozolomide for 8 weeks (2 cycles), in patients with retinoblastoma metastatic to the central nervous system (mass only) in two strata:

   * A. Initial diagnosis (mass)
   * B. At relapse (mass)
2. To determine hematologic toxicity: absolute neutrophil count (ANC), platelets and hemoglobin count.

Secondary Objectives:

1. To determine the response in other metastatic sites (non target) (orbit, bone marrow, bone, lung, liver and others)
2. To determine the remission rate and time to relapse on temozolomide.
3. To document the response of leptomeningeal metastasis (cerebrospinal fluid) to temozolomide

ELIGIBILITY:
Inclusion Criteria:

1. This study must be evaluated and confirmed by the local ethics committees and institutional review board of the participating institution, in accordance to the declaration of Helsinki. Informed consent must be administered and the parent or guardian must sign the document, authorized by the Ethics Committee and human subjects (therapy can not start if the documents are not signed).
2. Patients less than 21 years of age with diagnosis of retinoblastoma with metastasis to the CNS (central nervous system) must be confirmed by an ophthalmologist and/or a pathologist; in conjunction with the pediatric oncologist.
3. Metastasis to the CNS is defined as a mass in the chiasm or other site in the CNS, confirmed by MRI and/or

   CT:
   1. At diagnosis
   2. At relapse after conventional therapy.

   It is acceptable to have other sites of metastatic disease: lymphatic, bone, bone marrow or others.
4. All sites of metastasis must be measured in 3 planes, in millimeters and described in POND (Pediatric Oncology Network Database*)
5. Quality of life must be 3 by Lansky and 50% by Karnofksy
6. Hemogram: Hemoglobin of 7, ANC of 750, platelets of 75K.
7. Chemistry: direct bilirubin less than 3.0, indirect bilirubin less than 4.0, AST less 5x normal and ALT 5x normal, creatinine less than 1.5.
8. Treatment must start not more than 15 days from diagnosis of metastatic retinoblastoma.
9. Every patient with relapse or progression into the CNS must be documented with CT scan or MRI of the brain. Other sites of relapse may be evaluated, including bone marrow.
10. Patients who are newly diagnosed should have not received any other chemotherapeutic therapy (with the exception of dexamethasone) 1 week before starting, or radiotherapy, 4 weeks before starting.
11. All patients to be included in this study must be presented to the principal investigator using Horizon Live Web-conferencing through the Cure4Kids website. Eligibility and target CNS sites will be determined, as well as non-target sites.

Exclusion Criteria:

1. Patients with metastatic to CNS with only CSF involvement are NOT ELIGIBLE.
2. Relapse patients should have NOT received chemotherapy for 4 weeks, and no patient should have received nitroureas (melphalan, CCNU or mustard). No patient should have received radiation therapy in the previous 42 days. These patients are NOT eligible.
3. Diagnosis of AIDS or HIV positive.
4. Patients with disease NOT in the CNS are NOT eligible

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Response rate | 8 weeks
  Response rate (complete response plus partial response) of temozolomide for 8 weeks (2 cycles), in patients with retinoblastoma metastatic to the central nervous system (mass only) in two strata:
  1. Initial diagnosis (mass)
  2. At relapse (mass)
Evaluate the toxicity suffered during each cycle of temozolamide will be evaluated using the CTCAE v3.0 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Luna-Fineman, Principal Investigator — Stanford University
Locations (1):
- Unidad Nacional de Oncologia Pediatrica, Guatemala City, Guatemala